CLINICAL TRIAL: NCT01556646
Title: Effects of Tolvaptan on Cognitive Function, Brain Metabolism and Quality of Life in Hyponatremic Cirrhotics With Hepatic Encephalopathy: A Prospective Clinical Trial
Brief Title: Effect of Tolvaptan on Cognitive Function in Cirrhosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hunter Holmes Mcguire Veteran Affairs Medical Center (U.S. Federal Agency)
Collaborators: Otsuka America Pharmaceutical (Industry)
Responsible Party: Principal Investigator, Jasmohan Bajaj, Associate Professor of Medicine, Hunter Holmes Mcguire Veteran Affairs Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Bajaj 01720
Record Dates: First submitted 2012-03-15; First posted 2012-03-16 (Estimated); Last update posted 2014-02-07 (Estimated); Status verified 2014-02

CONDITIONS: Cirrhosis; Hepatic Encephalopathy; Hyponatremia
Keywords: Cirrhosis; Hepatic Encephalopathy; Hyponatremia; Brain MRI; Health-related quality of life; cognitive function
MeSH Terms: conditions — Fibrosis; Hepatic Encephalopathy; Hyponatremia | interventions — Tolvaptan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tolvaptan (Experimental): Open label study of tolvaptan. First 3 days as an inpatient then outpatient for the remainder of the study
  Interventions: Drug: Tolvaptan

INTERVENTIONS:
Drug: Tolvaptan — 15 to 30mg qd titrated to sodium concentration
  Other Names: Samsca

SUMMARY:
Hypothesis: Tolvaptan will improve cognitive function, brain edema and health-related quality of life in cirrhotic patients with hyponatremia

DETAILED DESCRIPTION:
Baseline assessment will include a

1. battery of eight cognitive tests
2. Health related quality of life
3. MRI head evaluating MR spectroscopy and diffusion tensor imaging

Patients will then be given tolvaptan 15-30mg qd for 14 days after which the tests will be repeated. During the first 3 days of tolvaptan administration, patients will be admitted and serum sodium will be drawn every 8 hours. 24 hr urine collection will also be performed.

Between the initiation and end of tolvaptan, patients will be seen at least every 3-5 days in between.

Participation will be terminated in case patients get transplanted or develop overt HE in between.

ELIGIBILITY:
Inclusion Criteria:

* Cirrhosis diagnosed by liver biopsy or radiological evidence of nodular cirrhotic liver or varices on endoscopy or laboratory features (platelet count <150,000 with an AST/ALT ratio >1).
* History of HE controlled on lactulose and/or rifaximin
* Last HE episode >2 months prior to enrollment and <2 episodes within 6 months
* Mini-mental status exam score ≥25
* Serum sodium <130mg/dl within the last 14 days and the day of enrollment
* Availability of a caregiver
* Able to undergo MR of the head

Exclusion Criteria:

* Uncontrolled HE manifested by MMSE <25
* Alcohol abuse within 3 months
* Illicit drug use within 3 months
* Psychoactive drug use other than regularly scheduled anti-depressants or methadone.
* Contraindication to MR examination (see attached MRI Safety Form)
* Placement of a transjugular intra-hepatic portosystemic shunt (TIPS)
* Creatinine Clearance less than 10 ml/min or undergoing hemodialysis
* HIV infection
* Use of azole medications
* Pregnancy
* Current use of tolvaptan, hypertonic saline or other medical therapies for hyponatremia

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2011-04; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Cognitive performance | 14 days

SECONDARY OUTCOMES:
Brain MR Spectroscopy | 14 days
Brain Diffusion Tensor Imaging | 14 days
Health-related Quality of Life | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Jasmohan S Bajaj, MD, Principal Investigator — Hunter Holmes McGuire VA Medical Center
Locations (1):
- Hunter Holmes McGuire VA Medical Center, Richmond, Virginia, United States